CLINICAL TRIAL: NCT00564707
Title: Comparison of Biofeedback Therapy and Botulinum Toxin Type A Injections for Treatment of Painful Levator Ani Syndrome in Women: A Randomized, Prospective Trial
Brief Title: Comparison of Biofeedback vs. Botox Injection to Treat Levator Ani Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 07-20034
Record Dates: First submitted 2007-11-26; First posted 2007-11-28 (Estimated); Last update posted 2007-11-28 (Estimated); Status verified 2007-11

CONDITIONS: Levator Ani Syndrome With Pain and/or Constipation Symptoms.
MeSH Terms: interventions — Biofeedback, Psychology; Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Standard biofeedback therapy will be given for painful levator ani syndrome over a course of eight weeks.
  Interventions: Behavioral: Biofeedback therapy
- 2 (Active Comparator): Botulinum toxin type A will be injected under EMG guidance into spastic and painful levator ani muscles. This may be repeated only twice on separate visits.
  Interventions: Procedure: Botulinum Toxin Type A Injection

INTERVENTIONS:
Behavioral: Biofeedback therapy — EMG guided biofeedback therapy using standard biofeedback computer software
  Arms: 1
Procedure: Botulinum Toxin Type A Injection — Under EMG guidance Botox is injected directly into the painful levator ani muscle.
  Arms: 2

SUMMARY:
Purpose: To assess whether EMG directed biofeedback therapy or Botulinum toxin type A injection of the levator ani muscles has any effect on pain from the levator ani syndrome, and, in addition, to what extent either treatment is superior to the other in terms of anorectal physiologic measurements, and quality of life.

Study Design: Randomized, prospective, unblinded double-armed study with crossover.

Methodology: Female subjects, aged 18 and over, with painful levator ani muscle spasm for at least one month duration will be randomized to receive either biofeedback therapy or Botulinum toxin type A injection. After randomization they will all undergo visual analog pain scoring, anorectal manometry, colonoscopy (if clinically indicated), and self-reported SF-36 quality of life measurement. Each patient will also complete numerical pain scale scoring, an SF-36, and a satisfaction questionnaire at each treatment visit and follow-up visit. Patients will submit these by mail. Identification numbers will be assigned to each subject for use on the SF-36 and Satisfaction Questionnaires throughout the study. Subjects will again undergo anorectal manometry at the end of their treatment arms. In the biofeedback arm patients will be treated biweekly for up to eight treatments and be provided exercises to practice at home based on their muscle function noted during the biofeedback training session. Subjects will keep a treatment diary of the exercises they do at home to help ensure compliance with the protocol. In the Botulinum toxin injection arm patients will be treated with scheduled injections of the levator ani muscles every six weeks for up to three total injections of 100U each. These injections will be directed to the painful areas of the levator muscles as guided by physical exam and EMG measurements. Should any patient fail their initial randomized treatment assignment (failure defined as "very dissatisfied" or "dissatisfied" on the satisfaction questionnaire), they will then be allowed to cross over to the other study arm. In addition to numerical pain scale scoring, an SF-36 questionnaire and anorectal manometry will also be repeated at the time of crossover. We intend to include all randomized patients in the final data analysis (according to their originally assigned treatment arm), regardless of outcome or reason for dropout, thus making this an "intent-to-treat" analysis.

Pivotal Study Definitions: The definition of adequate pain reduction, for the purposes of data analysis, will be a reduction in a subject's mean pain score of two on a numerical pain scale (0-10). Failure of either therapy will be defined as a response of "very dissatisfied" or "dissatisfied" on the satisfaction questionnaire at the end of either biofeedback (eight treatment visits) or Botulinum toxin (three injections) both before and after crossover.

Outcomes: We will determine the following for biofeedback therapy and Botulinum toxin type A injection: mean pain reduction, any differences in anorectal physiologic measurements (such as mean resting anal sphincter pressure), any changes in self-reported quality of life, and overall patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be 18 years of age or older and capable of providing informed consent indicating awareness of the investigational nature of this trial.
* History of chronic anorectal pain from levator ani spasm three or more months in duration.
* Pain involves only the anorectum, and is part of one of the established variants of levator ani syndrome including spasm, coccygodynia, proctalgia fugax.
* Written informed consent must be obtained from each patient prior to entering the study.
* Female patients will not be pregnant. Exclusion of the possibility of pregnancy by HCG testing (urine or serum) or by history (tubal ligation, hysterectomy, or menopause) is required prior to inclusion in the study.
* Patients should be willing to be followed within the military healthcare system during the course of study treatment and follow-up. Follow-up at other military facilities is acceptable.
* Ability to follow study instructions and likely to complete all required visits.

Exclusion Criteria:

* Patients with current participation in another clinical investigation of a medical device or a drug the requirements of which may preclude complete involvement in this study
* Active or previous (within 60 days prior to the study screening visit) chemotherapy
* Active or previous (within 60 days prior to the study screening visit) radiation
* Physical or mental disability or geographical concerns (residence not within reasonable travel distance) that would hamper compliance with required study visits
* The Investigator believes that the subject will be unwilling or unable to comply with study protocol requirements
* Patients < 18 years of age
* Incapable of providing informed consent
* Subject has chronic (>3 months) vaginal pain not related to levator spasm
* Patients who are pregnant.
* Patients unwilling, or unable, to be followed within the military healthcare system during the course of study treatment and follow-up.
* Documented urinary tract infection
* Genitourinary (GU) or anorectal malignancy
* Undergoing Botulinum toxin injection therapy or biofeedback therapy at the time of enrollment
* Known allergy or sensitivity to any study medication (Botulinum toxin, lidocaine)
* History of infection with Human Immunodeficiency Virus
* History of immunodeficiency disorders
* Patients taking antibiotics at the time of study enrollment
* Diagnosis of myasthenia gravis, Eaton-Lambert Syndrome, Amyotrophic Lateral Sclerosis, spinal cord injury or any other significant disease which might interfere with neuromuscular transmission.
* Concurrent use of agents that interfere with neuromuscular transmission
* Profound atrophy or excessive weakness on physical examination of the muscles to be injected with associated fecal incontinence
* Infection at the injection site
* Is overtly psychotic or suicidal.
* Anismus (inability to empty the rectum adequately during defecation) not associated with painful levator ani muscles
* History of anorectal or low pelvic surgery within the last year

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2007-08; Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Pain reduction from treatment with either Biofeedback, Botox injection, or both | Two years

SECONDARY OUTCOMES:
Anorectal physiologic changes - increase or decrease in anal sphincter pressures | Two years
Overall patient satisfaction | Two years
Patient quality of life | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery M Nelson, MD, Principal Investigator — Walter Reed Army Medical Center
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States